CLINICAL TRIAL: NCT00434200
Title: Interventional Study on the Effectiveness and Safety of Intensive Exercise in Patients With RA
Brief Title: Rheumatoid Arthritis Patients in Training
Acronym: RAPIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Health Care Insurance Board (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OG-97-024
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; exercise; damage
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

INTERVENTIONS:
Procedure: long-term intensive exercise

SUMMARY:
Aim of the study was to investigate the effectiveness (functional ability and physical capacity) and safety (disease activity and damage of the joints) of long-term high-intensity weight-bearing exercises in patients with rheumatoid arthritis (RA).The training proved to be safe and effective.

DETAILED DESCRIPTION:
The 300 patients with RA were randomized into two groups; exercise group and usual care group. The patients who participated in the 2 years intensive exercise training (2 times a week, training duration 65 minutes) improved their functional capacity and functional ability without detrimental effects on the large joints damage or on disease activity. Only patients with excessive large joint damage at baseline were at risk to develop additional damage when participating in intensive weight-bearing exercises. Patients who exercised were able to delay the decrease of bone mineral density of the hips.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis

Exclusion Criteria:

* Prosthesis of a weight bearing joint

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1998-01; Study Completion 2000-06

PRIMARY OUTCOMES:
effectiveness:
primary outcome:functional ability;MACTAR;6 months, 12 months, 18 months, 24 months
safety:
damage of the large joints (Larsen score); each year

SECONDARY OUTCOMES:
effectiveness:
muscle strength (strength of extensors of the knee); each 3 months and
aerobic fitness (ergometer); each 3 months
Safety:
disease activity (DAS) each 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Johanna MW Hazes, PhD, Principal Investigator — Erasmus Medical Centre

REFERENCES:
- [Background] de Jong Z, Munneke M, Zwinderman AH, Kroon HM, Ronday KH, Lems WF, Dijkmans BA, Breedveld FC, Vliet Vlieland TP, Hazes JM, Huizinga TW. Long term high intensity exercise and damage of small joints in rheumatoid arthritis. Ann Rheum Dis. 2004 Nov;63(11):1399-405. doi: 10.1136/ard.2003.015826. PMID 15479889
- [Background] de Jong Z, Munneke M, Jansen LM, Ronday K, van Schaardenburg DJ, Brand R, van den Ende CH, Vliet Vlieland TP, Zuijderduin WM, Hazes JM. Differences between participants and nonparticipants in an exercise trial for adults with rheumatoid arthritis. Arthritis Rheum. 2004 Aug 15;51(4):593-600. doi: 10.1002/art.20531. PMID 15334432
- [Background] de Jong Z, Munneke M, Lems WF, Zwinderman AH, Kroon HM, Pauwels EK, Jansen A, Ronday KH, Dijkmans BA, Breedveld FC, Vliet Vlieland TP, Hazes JM. Slowing of bone loss in patients with rheumatoid arthritis by long-term high-intensity exercise: results of a randomized, controlled trial. Arthritis Rheum. 2004 Apr;50(4):1066-76. doi: 10.1002/art.20117. PMID 15077288
- [Background] de Jong Z, Munneke M, Zwinderman AH, Kroon HM, Jansen A, Ronday KH, van Schaardenburg D, Dijkmans BA, Van den Ende CH, Breedveld FC, Vliet Vlieland TP, Hazes JM. Is a long-term high-intensity exercise program effective and safe in patients with rheumatoid arthritis? Results of a randomized controlled trial. Arthritis Rheum. 2003 Sep;48(9):2415-24. doi: 10.1002/art.11216. PMID 13130460